CLINICAL TRIAL: NCT05431049
Title: The Effect of Anesthesia Type on the Outcomes of Percutaneous Nephrolithotomy in Aging Male
Brief Title: Anesthesia Type on Percutaneous Nephrolithotomy in Aging Male
Status: Completed | Type: Observational
Sponsor: Sedat Önen (Other Government)
Collaborators: Bursa City Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Sedat Önen, Associate Professor, Bursa City Hospital
Organization: Bursa City Hospital (Other Government)
Other Study IDs: 2021-8/4
Record Dates: First submitted 2022-06-12; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Kidney Stone; Anesthesia
MeSH Terms: conditions — Kidney Calculi | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- combined spino-epidural anesthesia (CSEA): Percutaneous nephrolithotomy under combined spino-epidural anesthesia
  Interventions: Procedure: Percutaneous nephrolithotomy surgery (PNL)
- general anesthesia (GA): Percutaneous nephrolithotomy under general anesthesia
  Interventions: Procedure: Percutaneous nephrolithotomy surgery (PNL)

INTERVENTIONS:
Procedure: Percutaneous nephrolithotomy surgery (PNL) — Percutaneous nephrolithotomy (PNL) surgery was performed in all arms of the study to remove the renal stones. This surgery was performed with 2 anesthesia methods, CSEA and GA. These formed the groups of the study.
  Other Names: spino-epidural anesthesia (CSEA); general anesthesia (GA)

SUMMARY:
The aim of this study is to compare the anesthesia methods in percutaneous nephrolithotomy in terms of safety and effectiveness in elderly men.

DETAILED DESCRIPTION:
Data recorded since 2003 will be analyzed retrospectively. Elderly men with PNL will be divided into two groups according to the type of anesthesia. The results determined in both arms will be compared with appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Renal Stone Disease
* Above 65 years of age
* Male sex

Exclusion Criteria:

* Having low hemoglobin level before surgery
* Presence of hematology disease causing bleeding diathesis
* Presence of stones in an ectopic or transplanted kidney

Ages: 65 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Anesthesia results can differ, even with gender, due to pharmacokinetic reasons. Women are more resistant to general anesthesia and wake up earlier than men, and as a result, the time spent in an operating room was significantly shorter for women than for men.
  Because gender differences may affect the outcome of the study, we used male patients for whom we have the most data in our retrospective analysis.
Study Population: Above 65 years of age, male sex and having kidney stone
Sampling Method: Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Stone free rates | Post-surgery day 1
  These are the success percentages depending on the outcome of the surgical procedure in both groups.
Complication rates | During surgery to 24 hours after surgery
  These are the complication percentages depending on the outcome of the surgical procedure in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No